CLINICAL TRIAL: NCT06333197
Title: A Comparative Study Between the Retromandibular Transparotid Approach and Retromandibular Retroparotid Approach for Open Reduction and Internal Fixation of Mandibular Condylar Fracture.
Brief Title: Approaches for Open Reduction and Internal Fixation of Mandibular Condylar Fracture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa Mahmoud Hussien Ahmed, Resident doctor at general surgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mandibular condylar fracture
Record Dates: First submitted 2023-12-27; First posted 2024-03-27 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Mandibular Fractures
Keywords: Mandibular Condylar fracture; Approaches for mandibular fractures; Transparotid; Retromandibular; Comparative study; Retroparotid
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: ALL Patients diagnosed with Extra Capsular Fracture of Mandibular Condyle amenable for surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transparotid approch (Experimental): Patients who diagnosed with extra capsular fracture of mandibular condyle will undergo Retromandibular transparotid approch
  Interventions: Procedure: ORIF through transparotid approach
- Retroparotid approch (Experimental): Patients who diagnosed with extra capsular fracture of mandibular condyle will undergo Retromandibular retroparotid approch
  Interventions: Procedure: ORIF through retroparotid approach

INTERVENTIONS:
Procedure: ORIF through transparotid approach — The Retromandibular Transparotid approach is a surgical method used to access structures in the parotid gland region by making an incision behind the mandible.
  Arms: transparotid approch
Procedure: ORIF through retroparotid approach — The Retromandibular Retroparotid approach, also known as the Modified Blair Incision, is a surgical technique used to access structures within the parotid gland region by creating an incision behind the mandible and extending it into the parotid region.
  Other Names: ORIF through the Modified Blair Incision
  Arms: Retroparotid approch

SUMMARY:
The condylar region is the most frequent anatomical site for mandibular fractures .

Condylar fractures constitute 25.5% to 35.5% of all mandibular fractures. The mandibular condyle fracture is a type of fracture that affects the condyle, which is the knuckle-like projection of the mandible (lower jaw) that articulates with the temporal bone to form the temporomandibular joint (TMJ).

DETAILED DESCRIPTION:
Several approaches have been used for condylar fracture including intraoral, preauricular, submandibular and retromandibular approaches.

The selection of the appropriate surgical approach for condylar neck fracture represents a controversy.

The purpose of this Study is to Compare the outcomes and effectiveness between the retromandibular transparotid approach and retromandibular retroparotid approach for treatment of Condylar Fracture of Mandible.

ELIGIBILITY:
Inclusion Criteria:

* ALL Patients diagnosed with Extra Capsular Fracture of Mandibular Condyle amenable for surgery.

Exclusion Criteria:

* 1. Open Laceration in the condylar region. 2. Concomitant traumatic Facial Nerve injury. 3. Previous Surgery in Retromandibular region. 4. Severe Obese patients 5. Patients Refusing Surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Facial nerve injury | Up to 6 months
  Incidence of Facial Nerve Injury Following the Manoeuvre. ( Temporary or Permanent )
Operative time | Up to 3 hours
  The duration of the operation

SECONDARY OUTCOMES:
Fracture stability | Up to 3 Months
  Measure the status of bone after reduction
Mouth opening | Up to 3 Months
  Maximal inter incisor opening
Other Complication related to the Approach | Up to 6 Months
  Salivary Fistula, Sialocele, Freys Syndrome